CLINICAL TRIAL: NCT05562401
Title: Effect of Coconut Water Compared to Oral Electrolytes on Hydration Status in Adolescents Who Perform Physical Exercise: Randomized Clinical Trial, Double-blind
Brief Title: Effect of Coconut Water on Hydration Status in Pediatric Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Colima (Other)
Collaborators: Carmen Alicia Sanchez Ramirez (Unknown); Yunue Flores Ruelas (Unknown); Alexis Adan Lopez Maria (Unknown)
Responsible Party: Principal Investigator, Fabian Rojas Larios, Principal investigator, Universidad de Colima
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AALM
Record Dates: First submitted 2021-12-15; First posted 2022-09-30 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Sports Nutrition
Keywords: Dehydration; Pediatric population; Coconut water; Sport drink; Hydration status; Physical exercise
MeSH Terms: conditions — Dehydration; Motor Activity | interventions — Electrolytes

STUDY DESIGN:
Intervention Model Description: Two groups of subjects will be formed that will be randomized by the type of treatment they will receive, which will be the same during the 4 interventions of the study.
Who Masked: Participant, Investigator
Masking Description: The hydrating drinks will be placed in containers labeled as treatments 1 and 2 by a person in charge external to the project, where neither study subjects nor the main researcher will know the type of drink they will be receiving because both will have the same or similar appearance and taste.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coconut Water (Experimental): To determine if Coconut Water is more effective on hydration status than oral electrolytes in adolescents who perform physical exercise of aerobic competition.
  Interventions: Device: Coconut Water
- Oral Electrolytes (Active Comparator): To determine if Coconut Water is more effective on hydration status than oral electrolytes in adolescents who perform physical exercise of aerobic competition.
  Interventions: Drug: Oral Electrolytes

INTERVENTIONS:
Device: Coconut Water — Coconut water is the clear fluid inside the coconut, has natural electrolytes such as potassium, sodium and manganese.
  Arms: Coconut Water
Drug: Oral Electrolytes — Is be considered a drug that not require medical prescrption and containing water, carbohydrates and electrolytes.
  Arms: Oral Electrolytes

SUMMARY:
Introduction: The dehydration is a very common problem that is often not identified. The pediatric population is more susceptible to dehydration due to its physiological characteristics. Proper hydration is crucial for health since any degree of dehydration causes a reduction in physical and mental work capacity, hence the importance of preventing it by considering the type of drink. There are multiple beverage options, including industrial oral electrolytes (OE), on the other hand, coconut water (CW) has been studied as a natural alternative beverage with characteristics that can help maintain a state of euhydration. Objective: To determine if AC has a greater effect on hydration status than OE in adolescents who perform physical exercise. Material and methods: RCT, double blind. 34 subjects aged 13.02 ± 1.08 years were selected, assigned to treatment with either OE (Electrolit®) or CW. They received a weekly physical exercise session (4 weeks). Hydration was personalized (ml x kilograms of weight) and hydration was evaluated by Urine Specific Gravity (USG), Total Body Water (TBW) by bioimpedance and changes in body mass. Results:

Sesion 1 CW: Euhydrated (12) Dehydrated (5); OE: Euhydrated (8) Dehydrated (9); p value=0,16

Sesion 2 CW: Euhydrated (12) Dehydrated (5); OE: Euhydrated (7) Dehydrated (10); p value=0,08

Sesion 3 CW: Euhydrated (13) Dehydrated (4); OE: Euhydrated (13) Dehydrated (4); p value=1,00

Sesion 4 CW: Euhydrated (16) Dehydrated (1); OE: Euhydrated (8) Dehydrated (9); p value=0,007*

Conclusion: AC and OE have the same effect on hydration levels in adolescents who perform physical exercise.

DETAILED DESCRIPTION:
1. For current epidemiological reasons of Covid-19, an increase of 30% of losses has been considered already established in the sample size, giving a total of 22 participants per group (44 in total). For the same reason, two groups of 22 participants (11 experimental and 11 controls) will be divided in order to reduce the population and the risk of contagion, following the health protocols established by the institution mentioned in Annex 2. The type of randomization to be used in the study will be based on the assigned treatment (A / B) by the balanced block method. This method consists of assembling a series of blocks, made up of a certain number of cells, in which the different types of treatment are included. The number of blocks will be determined by the number of participants to be included and the number of cells that it has been decided to include in each block, so in the present study 12 blocks with four treatment cells will be placed, giving a total of 44 treatments to the same as the number of study subjects. Each block will contain in each cell one of the treatment alternatives and within each block there must be a balanced number of possible treatments. Treatments A and B will be written in blocks (22 with treatment A and 22 with treatment B). The randomization will be carried out by a person external to the study and the same person will be the one who will randomly assign the treatments in the blocks and the numbering of each block. They will be summoned to 12:00 noon on Monday or Tuesday only according to the group assigned to start with the collection of personal data (Annex 3) and a mental test called Psychological Characteristics related to Sports Performance (CPRD) (Annex 4) which will be applied by an expert in the area of psychology, in addition, if training is required for the application of the test, the main researcher will be trained to be able to perform it properly.
2. After taking personal data, hydrating drinks will be administered immediately before training (7 ml x kg of weight) 4 hours before. At 2:00 p.m., your corresponding hydrating drink (4 ml x kg of weight) will be administered again. Each participant will have a 600 ml graduated glass that will be granted by the researcher to keep track of the drink administered at the different times of each session.
3. Immediately afterwards, the anthropometry and urine sample will be taken. To record body mass, the protocol developed by the International Society for the Advancement of Kinanthropometry (ISAK) will be followed. The study subjects will be weighed in sports shorts and barefoot before starting physical exercise, having been told that, in the case of urinating or defecating, they should do so before the initial weigh-in. Simultaneously with taking the body mass, the% ACT will be determined by electrical bioimpedance. To record body mass and% of ACT water, the Tanita BC-533 bioimpedance scale will be used with a reliability of 97%, precision of 0.1kg and with a measuring range of 0-150kg.
4. Once the anthropometry and urine sample have been taken, a 200 ml dose will be administered immediately before exercise (10-15) min.
5. They will continue with the physical exercise protocol which will receive a physical exercise session per week (Tuesdays), with a duration of 1 hour and 15 minutes each session. The exercise sessions will be carried out in the Domingo Savio sports fields and will be taught by the principal investigator who has worked as a sports coach in the soccer area for 3 years, in addition to being trained for this purpose in the same institution where he was will carry out the study. Days prior to the start of the practical execution of the protocol, parents and selected students will be summoned to a meeting in order to explain the dynamics that will take place. The physical exercise sessions will consist of 4 parts:

   1. The first part of the workout will consist of a 10 minute warm-up and stretching to increase your basal HR and prepare the body for the next high intensity stages and prevent injuries in teens. The warm-up will have a break of 5 minutes and hydration of 2 ml x kg of weight.
   2. This second part will take place in 12 min of continuous jogging around the field at an average pace, aiming to do one lap every 1 minute 36 seconds, giving a total of 7 and a half laps to the soccer field (Cooper's Test). 8 min rest for the total recovery of energy systems and hydration of 2 ml x kg of weight.
   3. In the second part of the training, the adolescents must run from one line to another, twenty meters apart, at the pace set by a tape. This race pace will increase every minute. Subjects start the test at a speed of 8 km / hr, the first minute increases to 9 km / hr and thereafter, each minute increases the pace ½ km / hr. The test ends when they cannot keep up with the pace set (Test de course Navette). Approximate time 10 min with 8 min rest and hydration of 2 ml x kg of weight.
   4. In this last part of the training session, it is a type of exercise based on tabatas, which consists of performing 8 different exercises for 20 seconds per 10 seconds of rest to the rhythm of the marked music, giving a time of 4 minutes per tabata. .2 tabatas will be made with an intermediate rest of 3 min between each tabata and hydration of 2 ml x kg of weight.
6. At the end of this last stage of the training session, anthropometry and information collection will be taken where the percentage of weight change, body composition with bioimpedance will be determined before starting the final hydration, since if it is done at the In reverse, it is very likely that no one will come out in a state of dehydration. After the anthropometry, they will be administered the corresponding post-exercise hydration (1.5 ml x kg of weight) and the urine sample will be collected. In the event that a subject has not urinated due to dehydration, their sterilized bottle will be taken home and the head of research will be notified immediately for its proper conservation or transport.

   The calculation of the percentage of lost weight will be calculated using the following formula:% Weight Loss or Dehydration = [(Initial Weight - Final Weight) / Initial Weight] x 100.
7. As a final point, the data obtained before the exercise will be compared with the data obtained after the exercise, where the euhydration cut-off points will be analyzed to categorize the subject as dehydrated or euhydrated. An effective drink (CW or OE) will be considered when any 2 or more indicators (GEO, ACT or Body Mass) are consistent with the euhydration thresholds.

ELIGIBILITY:
Inclusion Criteria:

* Students that belong to "Instituto Salesiano Fray Pedro de Gante".
* Those students who are 12 years old and under 18 years of age.
* The parent or guardian of the adolescent and the student himself must agree to participate and comply with the autographed authorization of the informed consent letter.
* The adolescent must be in good physical and mental health.

Exclusion Criteria:

* Adolescents who suffer from a chronic disease such as obesity, hypertension, DM, asthma, COPD, cancer, injuries or physical disabilities.
* That the adolescent is allergic to any component of the treatments.

Elimination criteria:

* Adolescents who do not complete physical training sessions.
* That the adolescent presents a serious sports injury (fracture or sprain) during any of the physical exercise sessions.
* That the adolescent decides to withdraw once the practical research stage has begun.

Ages: 12 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: FABIAN ROJAS LARIOS, PhD, Study Director — frojas@ucol.mx; Carmen Alcia Sanchez Ramírez, PhD, Study Director — carmen_sanchez@ucol.mx
Locations (1):
- Alexis Adan Lopez Maria, Colima, Mexico

IPD SHARING:
Plan to Share IPD: No
At the moment there is the hesitation to share the information until having preliminary results.

REFERENCES:
- [Background] Saat M, Singh R, Sirisinghe RG, Nawawi M. Rehydration after exercise with fresh young coconut water, carbohydrate-electrolyte beverage and plain water. J Physiol Anthropol Appl Human Sci. 2002 Mar;21(2):93-104. doi: 10.2114/jpa.21.93. PMID 12056182
- [Background] Peart DJ, Hensby A, Shaw MP. Coconut Water Does Not Improve Markers of Hydration During Sub-maximal Exercise and Performance in a Subsequent Time Trial Compared with Water Alone. Int J Sport Nutr Exerc Metab. 2017 Jun;27(3):279-284. doi: 10.1123/ijsnem.2016-0121. Epub 2016 Oct 21. PMID 27768399

RESULTS

PARTICIPANT FLOW:
Recruitment Details: That the adolescent is a student belonging to the private institution ISFPG. That the adolescent perform competitive physical exercise of an aerobic type. Those students who are 12 years old and who are under 18 years old. The parent or guardian of the adolescent and the student himself must agree to participate and comply with The autograph authorization of the informed consent letter.
  The adolescent must be in good physical (Annex 2) and mental (Annex 3) health.
Pre-assignment Details: 34 healthy adolescents from 12 to 17 years of age were selected by simple sampling, of which 8 subjects were excluded due to CoVid-19 and 2 decided not to participate, later they were randomly assigned to a treatment group using the balanced block method.
Groups:
- Oral Electrolytes: To determine if Coconut Water is more effective on hydration status than oral electrolytes in adolescents who perform physical exercise of aerobic competition.
  OE: It is considered a medicine by the general health law that does not require a prescription and can be sold in any establishment that is not a pharmacy. Is an industrialized drink that containing water, carbohydrates, electrolytes.
Period: Overall Study
Arm/Group | Coconut Water | Oral Electrolytes
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Coconut Water: To determine if Coconut Water is more effective on hydration status than Oral Electrolytes in adolescents who perform aerobic physical exercise.
  Coconut Water: Coconut water is the clear fluid inside the coconut, has natural electrolytes such as potassium, sodium and manganese.
- Oral Electrolytes: To determine if Coconut Water is more effective on hydration status than Oral Electrolytes in adolescents who perform aerobic physical exercise.
  Oral electrolytes: It is considered a medicine by the general health law that does not require a prescription and can be sold in any establishment that is not a pharmacy.
- Total: Total of all reporting groups
Arm/Group | Coconut Water | Oral Electrolytes | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.06 (1.34) | 13 (0.79) | 13.03 (1.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 17 | 17 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: Kilograms] | 53.19 (10.85) | 61.82 (12.68) | 57.50 (12.42)
Height [Mean (Standard Deviation); unit: Centimeters] | 162.47 (11.81) | 162.53 (10.35) | 162.5 (10.93)

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Effect of AC vs EO on Hydration Status in Adolescents Who Perform Physical Exercise of Aerobic Competition.
Description: The independent variable is dichotomous and is classified as:
  A for coconut water and B for oral electrolytes. will be measured in milliliters.
  The dependient variable is dichotomus and is classified as:
  1. Euhydrated
  2. Dehydrated
  It will be classified as euhydrated or dehydrated when any 2 or more indicators are consistent with the euhydration or dehydration cut-off points, as the case may be.
Time Frame: 4 weeks
Measure: Number; unit: Number participants euhydrated
Arm/Group | Coconut Water | Oral Electrolytes
Number analyzed (Participants) | 68 | 68
Number participants euhydrated
  Ehuydrated | 53 | 36
  Dehydrated | 15 | 32

2. Secondary Outcome: Number of Participants With Dehydration Event After Exercise and Assigned Treatment Evaluated by Water Loss Related to Body Mass.
Description: The change in body mass will be measured in kg indicating dehydration in a loss equal to or greater than 5 percent of initial weight through the principle that 1g of weight lost is equivalent to 1ml of water lost.
Time Frame: 4 weeks
Reporting Status: Not Posted, anticipated posting 2024-12

3. Secondary Outcome: Number of Participants With a Dehydration Event After Exercise and the Assigned Treatment Evaluated by the Percentage of Water Lost by Bioelectrical Impedance.
Description: The electrical bioimpedance will measure the body water percentage before and after, indicating if the participant had the event of dehydration after the treatment when there was a loss of water equal to or greater than 2%.
Time Frame: 4 weeks
Reporting Status: Not Posted, anticipated posting 2024-12

4. Secondary Outcome: Number of Participants With Post-exercise Dehydration Event and Assigned Treatment Assessed by Urine Specific Gravity in g/Cubic cm.
Description: The level of light refraction in the urine of the subjects will be measured before exercise to ensure their state of euhydration and at the end the changes of the new urine sample will be seen post exercise and hydration. The specific gravity of urine will be expressed in g/cm3.
Time Frame: 4 weeks
Reporting Status: Not Posted, anticipated posting 2024-12

5. Secondary Outcome: Number of Participants With Post-exercise Dehydration Event in Both Assigned Treatments Assessed by Body Mass, Bioelectrical Impedance, and Urine Specific Gravity Using Chi-square or T-test.
Description: The results of each subject will be analyzed and both groups (coconut water or sports drink) will be compared to determine the hydration effect of the drinks used used by chi square or t tests.
Time Frame: 4 weeks
Reporting Status: Not Posted, anticipated posting 2024-12

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: The adverse event that could have occurred in addition to finishing the exercise session dehydrated would be: sports injury.
Arm/Group | Coconut Water | Oral Electrolytes
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
Some variables that could affect hydration levels and that, for economic reasons or beyond the control of the researchers in charge, could not be controlled or included in the study. The weather was an environmental factor that could not be controlled due to the facilities where the study was conducted. The gold standard of hydration was not applied for reasons of practicality and economy, in addition, hydration levels change in a matter of minutes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT05562401/Prot_SAP_ICF_001.pdf